CLINICAL TRIAL: NCT05402904
Title: Neurophysiological Assessment of Spinal Excitability in Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Kamel Khalaf, Principal Incestigator, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Soh-Med-22-05-05
Record Dates: First submitted 2022-05-15; First posted 2022-06-02 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Chronic Low-back Pain
MeSH Terms: interventions — Nerve Conduction Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with chronic low back pain (Active Comparator): 50 Patients will be recruited from neuropsychiatric outpatient clinic at Sohag University Hospital complaining of CLBP for more than 12 Weeks. Patients who are suspected of suffering from any autoimmune, rheumatological, or neurological disorders that could explain the pain that they experienced will be excluded from the study. Patients who are suffering from any disease that could affect the results and interpretation of the parameters of the H-reflex, F-wave or SSEP, including polyneuropathy and radiculopathy. Structural Spinal cause of pain will be excluded by relative investigations. Routine nerve conduction studies on both lower limbs as well as H-reflex, F-wave and SSEP will be performed on both patients and controls.Arabic versions of the Beck depression inventory and Taylor's Manifest Anxiety Scale will be used to measure depression and anxiety in both patients and healthy controls.
  Interventions: Diagnostic Test: nerve conduction study
- healthy controls (Active Comparator): 50 Healthy volunteers will be included in the control group of the study. Routine nerve conduction studies on both lower limbs as well as H-reflex, F-wave and SSEP will be performed on both patients and controls.
  Arabic versions of the Beck depression inventory and Taylor's Manifest Anxiety Scale (TMAS) will be used to measure depression and anxiety in both patients and healthy controls.
  Interventions: Diagnostic Test: nerve conduction study

INTERVENTIONS:
Diagnostic Test: nerve conduction study — Routine nerve conduction study on both lower limbs as well as F- wave , Hoffman reflex and somatosensory evoked potential.

SUMMARY:
Chronic low back pain (CLBP) is established by the persistence of low back pain beyond 3 months of symptom initiation . The overwhelming element of treatment is physical exercise . Other methods of treatment like cognitive therapy, behavioural therapy and multidisciplinary rehabilitation can also lead to significant improvements 1.

Prevalenc of CLBP increases linearly from the third decade of life on, until the 60 years of age, being more prevalent in women.2 CLBP is a common condition affecting many individuals at some point in their lives.3 The estimation is that between 5.0% and 10.0% of cases will develop CLBP, which is responsible for high treatment costs, sick leave, and individual suffering, in addition to being one of the main reasons for people to seek health care services.4 CLBP and related disorders represent a wide spectrum of syndromes that are associated with changes in the pain processing pathways of the central nervous system .5 Those syndromes affect many systems in the body, and the associated plasticity changes in the CNS can lead to augmentation of pain transmission and processing circuits. 6,7 The pain in patients with CLBP occurs as a result of a process called central sensitization (CS), which refers to increased excitability of the neurons in the dorsal horn of the spinal cord. This increased excitability is associated with increased spontaneous neuronal activity, expanded receptive fields, and enhanced responses to the impulses transmitted by both large and small-fiber sensory afferents.8 The Hoffman reflex , F-wave and Somatosensory evoked potential (SSEP) are often used to measure spinal excitability in various physiological and pathological states.9-10 The H-reflex is elicited by stimulation of type Ia afferent sensory fibers. These fibers synapse directly onto the alpha motor neurons in the anterior horn of the spinal cord, forming a monosynaptic reflex arc. Submaximal stimulation of this reflex arc elicits a compound muscle action potential (CMAP) known as the H wave. This reflex arc appears to depend on the balance between excitatory and inhibitory neurons in the spinal cord . F wave is a late response that follows the motor response (M) and is elicited by supramaximal electrical stimulation of a mixed or a motor nerve.11 The study of the F waves is particularly useful for the diagnosis of proximal nerve lesions that would be otherwise inaccessible to other routine NCSs.12 SSEPs are also important complementary diagnostic methods in the electrophysiologic evaluation of CLBP. SSEPs are a very sensitive measure of the functional integrity of the neuroaxis, including peripheral and central structures. When used in diagnostic mode they can provide additional information regarding the probable areas of dysfunction.

Since a change in spinal excitability is one of the main mechanisms underlying the hypothesis of CS in CLBP, performing these tests might be an easy, widely available, cheap, and objective method for assessing spinal excitability in patients with CLBP.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from chronic low back pain for more than 12 Weeks.

Exclusion Criteria:

1. Patients who are suspected of suffering from any autoimmune, rheumatological disorders that could explain the pain that they experienced will be excluded from the study.
2. Patients who are suffering from any disease that could affect the results and interpretation of the parameters of the H-reflex, F-wave or SSEP, including polyneuropathy and radiculopathy.
3. Patients who are suffering from any Structural Spinal cause of pain will be excluded by relative investigations.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Determine hoffman reflex latency in patient with chronic low back pain | 8 months
  Hoffman reflex latency will be measures in patient with chronic low back pain to assess spinal excitability
Determine F wave latency in patient with chronic low back pain | 8 months
  F wave latency will be measured in patient with chronic low back pain to assess spinal excitability

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Meucci RD, Fassa AG, Faria NM. Prevalence of chronic low back pain: systematic review. Rev Saude Publica. 2015;49:1. doi: 10.1590/S0034-8910.2015049005874. Epub 2015 Oct 20. PMID 26487293
- [Background] Knikou M, Murray LM. Repeated transspinal stimulation decreases soleus H-reflex excitability and restores spinal inhibition in human spinal cord injury. PLoS One. 2019 Sep 26;14(9):e0223135. doi: 10.1371/journal.pone.0223135. eCollection 2019. PMID 31557238
- [Background] Valat JP. Factors involved in progression to chronicity of mechanical low back pain. Joint Bone Spine. 2005 May;72(3):193-5. doi: 10.1016/j.jbspin.2004.07.010. No abstract available. PMID 15850987